CLINICAL TRIAL: NCT05399771
Title: Radiofrequency Hyperthermia Safety Study (RHySS)
Brief Title: Radiofrequency Hyperthermia Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: thermofield (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00075221
Record Dates: First submitted 2022-05-18; First posted 2022-06-01 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain; Soft Tissue Injuries; Wound Heal; Blood Flow
Keywords: mild hyperthermia
MeSH Terms: conditions — Chronic Pain; Soft Tissue Injuries | interventions — Laser-Doppler Flowmetry; Weights and Measures

STUDY DESIGN:
Intervention Model Description: 20 healthy subjects with intact skin on their lower legs that meet inclusion criteria - Participants will serve as their own control, by heating one leg and no the other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Thermofield temperature controlled radiofrequency device (Experimental): Participants will serve as their own control, by heating one leg and not the other. The radiofrequency device consists of a 4 by 6 inch heating pad connected to a temperature controller. The pad will be applied to the back of the leg and will covered using a compression stocking. The other leg will receive a pad and compression stocking, but radiofrequency will not be applied (no heating).
  Interventions: Device: Laser Doppler; Device: Radiofrequency Heating System; Device: Thermal Imaging; Other: Healthcare Questionnaire & Measurement

INTERVENTIONS:
Device: Laser Doppler — Study team will use a PeriScan PIM 3 System Laser Doppler to scan for blood perfusion before and after the Thermofield treatment. The PeriScan PIM 3 System is for non-invasive two-dimensional imaging of peripheral tissue.
  Other Names: PeriScan PIM 3 System Laser Doppler
Device: Radiofrequency Heating System — The radiofrequency will be set to achieve 42°C/107.6°F) and maintain this temperature consistently during the application time. This temperature is mild and may feel like a drugstore heating pad. The device will be turned on on one leg and will remain off on the other. The time for the heating will be 36 minutes, during which participants will remain in a reclined position, with their legs elevated. The device takes approximately 6 minutes to achieve a tissue temperature of 42°C, and the treatment time with consistent temperature application will be 30 minutes.
  Other Names: Thermofield
Device: Thermal Imaging — Study team will take thermal imaging photographs of the treatment area following each treatment.
Other: Healthcare Questionnaire & Measurement — A survey tool created to collect info from participants including:
  1. Name
  2. Age
  3. Weight/ height
  4. Pregnant or nursing?
  5. History of blood clots?
  6. Any wound healing problems?
  7. Any active open wounds on the legs?
  8. Any autoimmune disorders?
  9. Phone number
  10. Email address
  A measurement of the participants calf will be taken as well using a measuring tape.

SUMMARY:
This study will include 20 healthy subjects with intact skin on their lower legs that meet inclusion criteria. Participants will serve as their own control, by heating one leg and not the other. The radiofrequency device consists of a 4 by 6 inch heating pad connected to a temperature controller. Subjects will receive weekly treatments for 4 weeks, and will be re-evaluated 4 weeks after the last treatment to assess any tissue changes that continue after the treatments have concluded.

DETAILED DESCRIPTION:
This study will include 20 healthy subjects with intact skin on their lower legs that meet inclusion criteria below. Participants will serve as their own control, by heating one leg and not the other. The radiofrequency device consists of a 4 by 6 inch heating pad connected to a temperature controller. The pad will be applied to the back of the leg and will covered using a compression stocking. The other leg will receive a pad and compression stocking, but radiofrequency will not be applied (no heating).

At the first visit, subjects will be asked to fill out a healthcare questionnaire. With each weekly treatment, subjects will be evaluated to assess how their legs feel on a scale of 1-10, with 1 being no discomfort and 10 being intense pain. Their legs will be photographed before and after radiofrequency MH to examine any visible changes to the tissue. Study team will then use a PeriScan PIM 3 System Laser Doppler scanning for blood perfusion before the Thermofield treatment. The radiofrequency will be set to achieve 40°C/107.6°F) and maintain this temperature consistently during the application time. This temperature is mild and may feel like a drugstore heating pad. The device will be turned on on one leg and will remain off on the other. The time for the heating will be 36 minutes, during which participants will remain in a reclined position, with their legs elevated. The device takes approximately 6 minutes to achieve a tissue temperature of 40°C, and the treatment time with consistent temperature application will be 30 minutes. Study team will then use a PeriScan PIM 3 System Laser Doppler scanning for blood perfusion after the Thermofield treatment ends. Study team will take thermal imaging photographs of the treatment area following each treatment.

Subjects will receive weekly treatments for 4 weeks, and will be re-evaluated 4 weeks after the last treatment to assess any tissue changes that continue after the treatments have concluded. Subjects will be excluded from the study if they develop any kind of intolerance to the MH treatment, like increased pain or unexpected skin changes. If they receive a significant injury or wound that is not due to the study, such that the skin of the lower leg is no longer intact, they will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Healthy
* 20<BMI<40

Exclusion Criteria:

* Pregnant, nursing or child bearing potential
* Active infections of the skin in the lower leg
* Open or healing wounds on the lower leg
* Autoimmune disorder
* 40<BMI <20
* History of blood clots
* History of lower limb edema
* Tattoos and metal hardware in the leg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Levi, PhD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Legs
Period: Overall Study
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Started | 20; 40 Legs
Radiofrequency Heating System | 20; 20 Legs
No Heating | 20; 20 Legs
Completed | 16; 32 Legs
Not Completed | 4; 8 Legs
Not completed — Physician Decision | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Temperature Change- Skin Evaluation on Leg With Device
Description: To help determine safety during and after dermal application for generating elevated temperatures
Time Frame: week 1
Measure: Mean (Standard Error); unit: degrees
Units Other Than Participants: Legs
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 20
Number analyzed (Legs) | 20
degrees | 6.21 (0.478)

2. Primary Outcome: Mean Temperature Change- Skin Evaluation on Leg With Device
Description: To help determine safety during and after dermal application for generating elevated temperatures
Time Frame: week 2
Measure: Mean (Standard Error); unit: Degrees
Units Other Than Participants: legs
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 20
Number analyzed (legs) | 20
Degrees | 6.56 (0.63)

3. Primary Outcome: Mean Temperature Change- Skin Evaluation on Leg With Device
Description: To help determine safety during and after dermal application for generating elevated temperatures
Time Frame: week 3
Population: Subject 3 was withdrawn after treatment 2 because he developed a red spot and ultimately a small wound. Subject 9 and 10 were withdrawn after treatment 2 because they developed a lump under the skin.
Measure: Mean (Standard Error); unit: degrees
Units Other Than Participants: legs
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 17
Number analyzed (legs) | 17
degrees | 7.2 (0.67)

4. Primary Outcome: Mean Temperature Change- Skin Evaluation on Leg With Device
Description: To help determine safety during and after dermal application for generating elevated temperatures
Time Frame: week 4
Population: Subject 3 was withdrawn after treatment 2 - Subjects 9 and 10 were withdrawn after treatment 2 - Subject 8 did not complete - Subject 20 temperature check was not measured
Measure: Mean (Standard Error); unit: degrees
Units Other Than Participants: legs
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 15
Number analyzed (legs) | 15
degrees | 7.647 (0.62)

5. Primary Outcome: Mean Change in Blood Perfusion Assessment - mL/kg/Min
Description: Demonstrate that the Thermofield device improves blood flow to the tissue region where it has been applied.
  Laser Doppler scanning will be done on the skin before and after application of the hyperthermia device to quantitatively measure changes in blood perfusion after treatment. Blood perfusion via laser Doppler will also be used to asses increases or decreases in blood perfusion that would indicate harm, such as decreased perfusion - Blood flow is usually given in units mL/(100 g * min)
Time Frame: week 1
Population: change in pre and post perfusion for subjects at week 1 - Subject 3 was withdrawn
Measure: Mean (Standard Error); unit: mL/kg/min
Units Other Than Participants: legs
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 19
Number analyzed (legs) | 19
mL/kg/min | 430.312 (26.71)

6. Primary Outcome: Blood Perfusion Assessment - mL/kg/Min
Description: as for outcome 5
Time Frame: week 2
Population: change in pre and post perfusion for subjects at week 2 - Subject 3 was withdrawn
Measure: Mean (Standard Error); unit: mL/kg/min
Units Other Than Participants: legs
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 19
Number analyzed (legs) | 19
mL/kg/min | 414.065 (30.77)

7. Primary Outcome: Blood Perfusion Assessment - mL/kg/Min
Description: as for outcome 5
Time Frame: week 3
Population: change in pre and post perfusion for subjects at week 3 - Subject 3 was withdrawn after treatment 2 - Subjects 9 and 10 were withdrawn after treatment 2
Measure: Mean (Standard Error); unit: mL/kg/min
Units Other Than Participants: legs
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 17
Number analyzed (legs) | 17
mL/kg/min | 470.147 (37.85)

8. Primary Outcome: Blood Perfusion Assessment - mL/kg/Min
Description: as for outcome 5
Time Frame: week 4
Population: change in pre and post perfusion for subjects at week 4 - Subject 3 was withdrawn after treatment 2 - Subjects 9 and 10 were withdrawn after treatment 2 - Subject 8 did not complete - Subject 16 perfusion check was not measured
Measure: Mean (Standard Error); unit: mL/kg/min
Units Other Than Participants: legs
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 15
Number analyzed (legs) | 15
mL/kg/min | 434.967 (31.96)

9. Primary Outcome: Blood Perfusion Assessment - mL/kg/Min
Description: as for outcome 5
Time Frame: week 8
Population: Perfusion without treatment at week 8 - Subject 3 was withdrawn after treatment 2 - Subjects 9 and 10 were withdrawn after treatment 2 - Subject 8 did not complete
Measure: Mean (Standard Error); unit: mL/kg/min
Units Other Than Participants: legs
Groups:
- Thermofield Temperature Controlled Radiofrequency Device: Participants will serve as their own control. No Thermofield treatment at week 8.
  Laser Doppler: Study team will use a PeriScan PIM 3 System Laser Doppler to scan for blood perfusion before and after the Thermofield treatment. The PeriScan PIM 3 System is for non-invasive two-dimensional imaging of peripheral tissue.
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 16
Number analyzed (legs) | 16
mL/kg/min | 29.659 (1.68)

10. Primary Outcome: Change in Comfort Level Scores of Participants Receiving Hyperthermia Treatment
Description: A pain score/ 'How are you feeling?' survey will be used at each session before and after hyperthermia treatment. The scale of 0 meaning non pain/ feel fine to 10 being the maximum pain/ not feeling well will be used.
Time Frame: week 1
Population: Subject 3 was withdrawn
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Thermofield Temperature Controlled Radiofrequency Device: Participants will serve as their own control, by heating one leg and not the other. The radiofrequency device consists of a 4 by 6 inch heating pad connected to a temperature controller. The pad will be applied to the back of the leg and will covered using a compression stocking. The other leg will receive a pad and compression stocking, but radiofrequency will not be applied (no heating).
  Laser Doppler: Study team will use a PeriScan PIM 3 System Laser Doppler to scan for blood perfusion before and after the Thermofield treatment. The PeriScan PIM 3 System is for non-invasive two-dimensional imaging of peripheral tissue.
  Radiofrequency Heating System: The radiofrequency will be set to achieve 42°C/107.6°F) and maintain this temperature consistently during the application time. This temperature is mild and may feel like a drugstore heating pad. The device will be turned on on one leg and will remain off on the other. The time for the heating will be 36 minutes, during which participants will remain in a reclined position, with their legs elevated. The device takes approximately 6 minutes to achieve a tissue temperature of 42°C, and the treatment time with consistent temperature application will be 30 minutes.
  Patients will be asked to rate their pain pre and post thermofield treatment on a scale from 0-10, with o being no pain and 10 being the worst pain imaginable.
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 19
score on a scale | 0.1 (0.10)

11. Primary Outcome: Change in Comfort Level Scores of Participants Receiving Hyperthermia Treatment
Description: as for outcome 10
Time Frame: week 2
Population: Subject 3 was withdrawn
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 19
score on a scale | 0.21 (0.14)

12. Primary Outcome: Change in Comfort Level Scores of Participants Receiving Hyperthermia Treatment
Description: as for outcome 10
Time Frame: week 3
Population: Subject 3 was withdrawn after treatment 2 - Subjects 9 and 10 were withdrawn after treatment 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 17
score on a scale | 0.176 (0.09)

13. Primary Outcome: Change in Comfort Level Scores of Participants Receiving Hyperthermia Treatment
Description: as for outcome 10
Time Frame: week 4
Population: Subject 3 was withdrawn after treatment 2 - Subjects 9 and 10 were withdrawn after treatment 2 - Subject 8 did not complete
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 16
score on a scale | 0.375 (0.20)

14. Primary Outcome: Change in Comfort Level Scores of Participants Receiving Hyperthermia Treatment
Description: as for outcome 10
Time Frame: week 8
Population: as for outcome 13
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 16
score on a scale | 0 (0)

15. Primary Outcome: Safety: Number of Blister Formations
Description: Cumulative number of blisters formed across all participants during weekly sessions from week 1 to 8 is reported in the data table.
Time Frame: From week 1 through week 8
Measure: Number; unit: blisters observed
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 20
blisters observed | 0

16. Primary Outcome: Safety: Significant Changes in Redness
Description: Number of participants with significant changes in redness that required intervention.
Time Frame: from week 1 through week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 20
Participants | 0

17. Secondary Outcome: Number of Participants Who Attended the Session
Description: The number of participants who attend hyperthermia sessions will be documented.
Time Frame: week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 20
Participants | 20

18. Secondary Outcome: Number of Participants Who Attended the Session
Description: The number of participants who attend hyperthermia sessions will be documented.
Time Frame: week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 20
Participants | 20

19. Secondary Outcome: Number of Participants Who Attended the Session
Description: The number of participants who attend hyperthermia sessions will be documented.
Time Frame: week 3
Population: Subject 3 was withdrawn after treatment 2 - Subjects 9 and 10 were withdrawn after treatment 2
Measure: Count of Participants; unit: Participants
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 17
Participants | 17

20. Secondary Outcome: Number of Participants Who Attended the Session
Description: The number of participants who attend hyperthermia sessions will be documented.
Time Frame: week 4
Population: Subject 8 did not complete this visit
Measure: Count of Participants; unit: Participants
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
Number analyzed (Participants) | 17
Participants | 16

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the life of the study (8 weeks).
Arm/Group | Thermofield Temperature Controlled Radiofrequency Device
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thermofield Temperature Controlled Radiofrequency Device (N=20)
Burn/knot (Skin and subcutaneous tissue disorders) | 3 (3) — 1 Subject experienced superficial burn and 2 others experienced a tender "knot" under the skin where the heating pad had been placed (L calf). All 3 Subjects were WD from the study and followed until healed. All 3 received therapeutic radiofrequency

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT05399771/Prot_SAP_003.pdf
  • Informed Consent Form (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT05399771/ICF_002.pdf